CLINICAL TRIAL: NCT04845568
Title: Testing Digital Technologies to Help Families Build Healthy Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202004074
Record Dates: First submitted 2021-03-03; First posted 2021-04-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Childhood Obesity
Keywords: Virtual Reality; Obesity; Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: Participants are randomized to control or intervention. The control condition is watching a video and playing a brief computer game, while the intervention condition consists of the virtual reality experience. Each provides child-friendly nutrition education as well as education on consideration of future consequences.
Masking Description: No masking. Outcomes will be assessed via surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (No Intervention): This is the control condition, which views a short video and online interactive game with psychoeducational material on healthy eating and consideration of future consequences.
- Virtual Reality (Experimental): This is the intervention condition, which participates in the virtual reality experience; the experience includes psychoeducational material on healthy eating and consideration of future consequences.
  Interventions: Behavioral: Virtual Reality Experience

INTERVENTIONS:
Behavioral: Virtual Reality Experience — The virtual reality experience includes psychoeducation content about healthy eating and consideration of future consequences. It includes a game where participants are in a go kart and pick up healthy or unhealthy foods on the road. Participants play in the "present" and in the "future."
  Arms: Virtual Reality

SUMMARY:
The current study is a randomized pilot trial to test the feasibility of a psychoeducational virtual reality experience to increase motivation for behavior change among children with overweight or obesity.

DETAILED DESCRIPTION:
The investigators will be conducting a randomized pilot trial to compare a virtual reality (VR) experience to a video. Each provides child-friendly nutrition education as well as education on consideration of future consequences (episodic future thinking). The video acts as the control condition such that we might begin to understand whether the psychological presence produced by virtual reality might increase motivation for behavior change.

The VR experience consists of a game in which participants play a racing game collecting healthy or unhealthy foods on the road. Collection of healthy foods increases speed, and collection of unhealthy foods decreases speed. Participants then play in the "future" where the food choices they made in the past also affect how they can move in the future game. If they collected mostly unhealthy foods in the past they move slower in the future, and if they collected healthy foods in the past they move faster in the future. However, foods collected in the future game can also change their speed, and participants are able to experience both future conditions i.e. they play in the future condition depending on if they ate healthily or not in the past, and then they play in the opposite future condition. A narrator in the game provides information on making healthy choices and about considering future consequences. The control video covers similar education on making healthy choices and considering future consequences. Additionally, the control video condition also includes a short computer-based game about healthy eating.

The investigators will enroll 60 English-speaking children ages 6-12 with overweight or obesity who are not in behavioral treatment to address weight and one of their parents. Participants will be recruited from the community using methods such as social media and flyers and will complete a phone-screen to determine initial eligibility. Participants determined to be eligible over the phone will come for an in-lab visit. In-lab, children will provide verbal assent and parents provide written informed consent. Children and parents will complete baseline measures, including having height and weight taken, demographic survey questions, assessment of participants' eating and physical activity behaviors, and other survey assessments selected to evaluate participants' behavioral beliefs, behavioral intentions, affect, and motivation for behavior change. Post-video or -VR participants will take the same survey assessments aimed at evaluating behavioral beliefs, intentions, affect and motivation for behavior change. Additionally, all participants will take usability assessments to determine the acceptability of the video or VR and participants randomized to the VR will complete measures to evaluate how immersive the VR seemed. At 2-week follow-up participants will again report their eating and physical activity behaviors and some cognitive measures in order to see whether the VR may have impacted behavior and cognitions.

ELIGIBILITY:
This study is enrolling guardian and child dyads.

Eligibility criteria include:

1. Parent is biological or legal guardian and can therefore consent on behalf of the child
2. Parent is under 80 years old and child is between 6 and 12 years old
3. Child BMI is at or above the 85th percentile for age and sex
4. Parent BMI is at or above 25

Exclusion Criteria include:

1. Child is in behavioral weight-loss treatment (behavior weight-loss treatment will not include if their pediatrician is counseling them on their weight, but instead refers to intensive outpatient behavioral treatment for overweight/obesity only) 6. Child or parent have a history of seizures, a history of severe psychiatric conditions such as Schizophrenia or Paranoia, or use any medical devices such as pacemakers 7. Child is exhibiting any disordered eating behavior (i.e. purging, laxative or diuretic use)

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Fitzsimmons-Craft, PhD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Consent to share data is collected and available upon reasonable request after the publication of main outcomes.

REFERENCES:
- [Derived] Fowler LA, Vazquez MM, DePietro B, Wilfley DE, Fitzsimmons-Craft EE. Development, usability, and preliminary efficacy of a virtual reality experience to promote healthy lifestyle behaviors in children: pilot randomized controlled trial. Mhealth. 2024 Oct 21;10:29. doi: 10.21037/mhealth-24-24. eCollection 2024. PMID 39534453

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video | Virtual Reality
Started | 26 (These are the total number of unique children (n=13) and caregivers (n=13) that started the study (13 children + 13 caregivers = 26 unique participants).) | 28 (These are the total number of unique children (n=14) and caregivers (n=14) that started the study (14 children + 14 caregivers = 28 unique participants).)
Completed | 26 (These are the total number of unique children (n=13) and caregivers (n=13) that completed the study (13 children + 13 caregivers = 26 unique participants).) | 28 (These are the total number of unique children (n=14) and caregivers (n=14) that completed the study (14 children + 14 caregivers = 28 unique participants).)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Children and caregivers were randomly assigned to either the control (video) or the virtual reality arm. Assignments to condition happened as a pair. For reporting purposes, two separate arms represent children and caregivers for each condition.
Groups:
- Video (Children); Video (Caregivers): This is the control condition, which views a short video and online interactive game with psychoeducational material on healthy eating and consideration of future consequences.
- Virtual Reality (Children); Virtual Reality (Caregivers): This is the intervention condition, which participates in the virtual reality experience; the experience includes psychoeducational material on healthy eating and consideration of future consequences.
  Virtual Reality Experience: The virtual reality experience includes psychoeducation content about healthy eating and consideration of future consequences. It includes a game where participants are in a go kart and pick up healthy or unhealthy foods on the road. Participants play in the "present" and in the "future."
- Total: Total of all reporting groups
Arm/Group | Video (Children) | Virtual Reality (Children) | Video (Caregivers) | Virtual Reality (Caregivers) | Total
Number analyzed (Participants) | 13 | 14 | 13 | 14 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.02 (2.21) | 10.66 (1.51) | 45.31 (6.07) | 43.71 (8.29) | 27.43 (19.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 10 | 12 | 36
  Male | 7 | 6 | 3 | 2 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 0 | 4
  Not Hispanic or Latino | 11 | 14 | 11 | 14 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 2 | 4 | 13
  White | 9 | 7 | 10 | 9 | 35
  More than one race | 2 | 1 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 | 13 | 14 | 54

OUTCOME MEASURES:

1. Primary Outcome: Acceptability as Measured by the System Usability Scale
Description: The System Usability Scale (SUS) was used to measure usability of the intervention. The items were adapted so that the caregiver could report on their child's experience of usability. SUS consists of 10 items with five response options on a Likert scale: strongly disagree (0) to strongly agree (4). SUS yields a single number representing a composite measure of the overall usability of a system being studied, ranging from 1 to 100, with greater scores reflecting greater usability, and calculated as follows (Brooke, 1996): "Each item's score contribution will range from 0 to 4. For items 1,3,5,7,and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. Multiply the sum of the scores by 2.5 to obtain the overall score."
Time Frame: Assessed immediately after the 10-minute, single-session, in-person virtual reality or video intervention
Population: Data were reported by the caregivers, who reported for both the child and themselves. Only one score is reported for each child-caregiver dyad.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
scores on a scale | 80.63 (10.72) | 76.54 (17.66)

2. Primary Outcome: Acceptability as Measured by the Usefulness, Satisfaction and Ease of Use Questionnaire
Description: The Usefulness, Satisfaction and Ease of Use Questionnaire was used to measure acceptability, specifically usefulness, ease of use, ease of learning, and satisfaction with an intervention or service. Items were adapted to have the caregivers report on their child's experience of usability. The shortened instrument used in this study (Lund, 2001) contains 19 items, and respondents indicate their agreement with each statement on a scale from 1 (strongly disagree) to 7 (strongly agree). Scores are summed to create an overall score of usability, ranging from 19 to 133, with greater scores indicating greater usability.
Time Frame: Assessed immediately after the 10-minute, single-session, in-person virtual reality or video intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
score on a scale | 75.58 (12.67) | 79.31 (15.67)

3. Primary Outcome: Acceptability as Measured by Degree of Immersion (for Those in the Virtual Reality Condition)
Description: Degree of Immersion in the virtual environment is assessed by parent self-report with the Presence Questionnaire (Witmer 2005). The Presence Questionnaire is a 24 item questionnaire that assesses involvement, auditory fidelity, adaption/immersion, interface quality, consistency with expectations, and haptic/visual fidelity. Given that sense of touch was not applicable to the present study, this item (23) was not included in the final score. Responses to the items are on a scale from 1 (not at all) to 7 (completely), and responses are summed to create an overall score. Potential scores range from 23 to 161, with greater scores indicating greater self-reported feelings of being immersed in the virtual environment.
Time Frame: Assessed immediately after the 10-minute, single-session, in-person virtual reality intervention
Population: Data were collected in Virtual Reality condition only. Data were reported by the caregivers, who reported for both the child and themselves. Only one score is reported for each child-caregiver dyad.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 0 | 14
score on a scale |  | 116.92 (20.22)

4. Primary Outcome: Acceptability as Measured by Child Interview Questions
Description: Assessed with child interview questions created by the study team. Questions ask children to respond by indicating which smiley face on a 5 point analog scale best represents how they feel, from 1 (unhappy/not at all) to 5 (very happy/a lot). Acceptability was assessed by asking how much the child liked the intervention, and motivation was assessed by asking the child how motivated they are to eat healthier post-intervention. Greater numbers on each question represent greater acceptability and greater post-intervention motivation, respectively.
Time Frame: Assessed immediately after the 10-minute, single-session, in-person virtual reality or video intervention
Population: Data were reported by the child only. This item was not collected from caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
score on a scale
  Acceptability (1 question) | 3.54 (0.84) | 4.31 (0.48)
  Motivating (1 question) | 4.08 (1.00) | 3.69 (.86)

5. Primary Outcome: Change in Self-Efficacy for Healthy Eating and Physical Activity (SE-HEPA)
Description: Child self-report survey measure. The Self-Efficacy for Healthy Eating and Physical Activity (SE-HEPA) measure was developed by Steele, Bindler, Power, and Daratha (2008) and is based on Motl et al.'s (2000) unidimensional measure of self-efficacy for exercise. Based on Bandura's (1977) social cognitive theory, SE-HEPA was designed to evaluate a children's or adolescents' confidence in their ability to engage in healthy eating (8 items) and physical activity behaviors (8 items). Items are answered on 5 point Likert scales from strongly disagree (1) to strongly agree (5). Scores are summed to create two subscales: self-efficacy for healthy eating, and self-efficacy for physical activity. Possible scores for each subscale range from 8 to 40, with greater scores indicating greater self-efficacy.
Time Frame: Assessed at baseline (before the intervention) and immediately after the 10-minute, single-session, in-person virtual reality or video intervention
Population: Data were reported by the child only. These data were not collected from caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
score on a scale
  Pre-intervention healthy eating | 26.08 (9.68) | 26.64 (6.87)
  Post-intervention healthy eating | 28.69 (9.89) | 28.07 (7.89)
  Pre-intervention Physical Activity | 24.08 (7.32) | 23.64 (8.05)
  Post-intervention Physical Activity | 26.23 (9.37) | 26.93 (7.73)
Statistical Analysis 1: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in Self-Efficacy for Physical Activity. It is an independent samples t test. It is testing the null hypothesis that the mean change in self-efficacy for physical activity does not differ between conditions; Test type: Superiority; p = 0.592, t-test, 2 sided — A priori threshold for statistical significance was set at p<0.05; Degrees of freedom = 25; Mean Difference (Net) = 1.13, 95% CI 2-sided [-3.16 to 5.43], Standard Error of Mean 2.08
Statistical Analysis 2: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in Self-Efficacy for Healthy Eating. It is an independent samples t test. It is testing the null hypothesis that the mean change in self-efficacy for healthy eating does not differ between conditions; Test type: Superiority; p = 0.453, t-test, 2 sided — A priori threshold for statistical significance was set at p<0.05; Degrees of freedom = 25; Mean Difference (Net) = -1.19, 95% CI 2-sided [-4.39 to 2.02], Standard Error of Mean 1.56

6. Primary Outcome: Change in Caregiver Readiness to Change Diet and Physical Activity
Description: The caregiver Readiness to Change Diet and Physical Activity items were adapted from previously used questions and designed to assess caregiver readiness to help their child change physical activity and eating behaviors. Parents self-report their intentions to help their children with healthy habits by answering "Do you intend to find ways to improve the way your child eats?" and "Do you intend to find ways to improve your child's physical activity level?" with responses from 1 ("No, and I'm not intending to make changes"), 2 ("Yes, I intend to make changes in the next 6 months"), 3 ("Yes, I intend to make changes in the next month"), to 4 ("I'm already helping my child improve their [eating/activity]"). Scores range from 1 to 4, with greater scores indicating greater caregiver readiness to help their child change. Items are not aggregated, and each item is analyzed separately.
Time Frame: Items are assessed immediately pre intervention and at 2-weeks after intervention
Population: Data were reported by the caregivers only. Only one score is reported for each child-caregiver dyad. These measures were not collected from children.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
score on a scale
  Pre-intervention intend to help child change eating | 3.15 (.80) | 3.43 (.51)
  Two-week post-intervention intend to help child change eating | 3.31 (.86) | 3.86 (.36)
  Pre-intervention intend to help child change activity | 3.08 (.86) | 3.29 (.73)
  Two-week Post-intervention intend to help child change activity | 3.31 (.95) | 3.64 (.63)
Statistical Analysis 1: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in Caregiver Readiness to Change Child's Eating. It is an independent samples t test. It is testing the null hypothesis that the mean change in readiness for healthy eating does not differ between conditions; Test type: Superiority; p = .368, t-test, 2 sided — A priori threshold for statistical significance set at p< 0.05; Degrees of freedom = 25; Mean Difference (Net) = 0.275, 95% CI 2-sided [-.342 to .892], Standard Error of Mean .300
Statistical Analysis 2: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in Caregiver Readiness for Physical Activity. It is an independent samples t test. It is testing the null hypothesis that the mean change in caregiver intentions to help child improve physical activity from baseline to two-week follow up does not differ between conditions; Test type: Superiority; p = .714, t-test, 2 sided — A priori threshold for statistical significance set at p< .05; Degrees of freedom = 25; Mean Difference (Net) = .126, 95% CI 2-sided [-.575 to .827], Standard Error of Mean .340

7. Primary Outcome: Change in Behavioral Beliefs (Attitudes) and Intentions
Description: Behavioral beliefs (attitudes) and intentions toward health eating were measured with items adapted from previous literature based on the Theory of Planned Behavior. Where needed, language was adapted to lower the reading level for child participants. Items were answered on 7 point Likert scales from strongly disagree (1) to strongly agree (7). Scores were summed for child attitudes (beliefs), child intentions, and caregiver intentions, self-reported by children and caregivers pre- and post-intervention. Eight items measured child attitudes towards eating healthy, with total scores ranging from 8 to 56, and greater scores indicating more positive attitudes toward eating healthier.
  Six items measured child intentions toward healthy eating, with total scores ranging 6 to 42, and greater scores indicating greater intentions to engage in the behavior.
  Four items measured caregiver intentions to help child, with total scores ranging from 4 to 28, and greater scores indicating gre
Time Frame: At baseline and after the 10-minute, single-session, in-person intervention
Population: The outcome measures were analyzed separately for children and caregivers. Data below was collected by either the child only or the caregiver only, as indicated in the row title. Different measures were collected for children and caregivers, as indicated in the measure description.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
score on a scale
  Pre-Intervention Child Intentions toward healthy eating | 27.62 (10.74) | 25.14 (9.45)
  Post-Intervention Child Intentions toward healthy eating | 31.46 (11.10) | 27 (8.8)
  Pre-Intervention Child attitudes toward healthy eating | 21.31 (7.18) | 19.36 (4.13)
  Post-Intervention Child Healthy eating attitudes | 21.85 (7.12) | 21.71 (5.01)
  Pre-Intervention parent intentions toward healthy eating | 24.54 (3.13) | 24.36 (6.28)
  Post-Intervention parent intentions toward healthy eating | 25 (3.14) | 26.93 (1.94)
Statistical Analysis 1: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child attitudes toward healthy eating. It is an independent samples t test. It is testing the null hypothesis that the mean change in child attitudes toward healthy eating from baseline to post-intervention does not differ between conditions; Test type: Superiority; p = .783, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = -.522, 95% CI 2-sided [-4.39 to 3.34], Standard Error of Mean 1.88
Statistical Analysis 2: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child intentions toward healthy eating. It is an independent samples t test. It is testing the null hypothesis that the mean change in child intentions toward healthy eating from baseline to post-intervention does not differ between conditions; Test type: Superiority; p = .323, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = -1.99, 95% CI 2-sided [-6.05 to 2.07], Standard Error of Mean 1.97
Statistical Analysis 3: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in caregiver intentions toward helping their child engage in healthy eating. It is an independent samples t test. It is testing the null hypothesis that the mean change in caregiver intentions from baseline to post-intervention does not differ between conditions; Test type: Superiority; p = .276, t-test, 2 sided — A priori threshold for statistical significance is set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = 2.11, 95% CI 2-sided [-1.79 to 6.01], Standard Error of Mean 1.89

8. Secondary Outcome: Change in Child Diet
Description: Parents reported on their child's eating behavior of the previous week with three different items asking parents to report the number of servings per week the child ate of fruits, vegetables, and fast foods.
Time Frame: Immediately pre intervention/control and at 2 week follow-up
Population: Data were reported by the caregivers, who reported for on the child's behavior. Only one score is reported for each child-caregiver dyad.
Measure: Mean (Standard Deviation); unit: servings per week
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
servings per week
  Pre-intervention Weekly intake of fruits | 3.23 (1.42) | 3.50 (1.09)
  Pre-intervention Weekly intake of vegetables | 2.85 (.9) | 3.5 (.86)
  Pre-intervention Weekly intake of fast foods | 2 (.58) | 2.14 (1.1)
  Two-week Post-intervention Weekly intake of fruits | 2.77 (1.30) | 3.29 (1.07)
  Two-week Post-intervention Weekly intake of vegetables | 2.92 (1.12) | 3.57 (0.94)
  Two-week Post-intervention Weekly intake of fast food | 1.85 (.56) | 1.79 (.7)
Statistical Analysis 1: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child intake of fruits. It is an independent samples t test. It is testing the null hypothesis that the mean change in child fruit servings per week from baseline to two-week follow up does not differ between conditions; Test type: Superiority; p = .547, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = .247, 95% CI 2-sided [-.59 to 1.08], Standard Error of Mean .40
Statistical Analysis 2: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child intake of vegetables. It is an independent samples t test. It is testing the null hypothesis that the mean change in child vegetable servings per week from baseline to two-week follow up does not differ between conditions; Test type: Superiority; p = .990, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = -.005, 95% CI 2-sided [-.87 to .86], Standard Error of Mean .42
Statistical Analysis 3: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child intake of fast food. It is an independent samples t test. It is testing the null hypothesis that the mean change in child fast food servings per week from baseline to two-week follow up does not differ between conditions; Test type: Superiority; p = .527, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = -.203, 95% CI 2-sided [-.86 to .45], Standard Error of Mean .32

9. Secondary Outcome: Change in Child Eating Behavior
Description: Parents reported on their child's eating behavior of the previous week with two different items asking parents to report the number of days per week the child ate breakfast and family dinner.
Time Frame: Immediately pre intervention/control and at 2 week follow-up
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
days per week
  Pre-intervention family dinner | 4.54 (2.11) | 4.93 (2.50)
  Pre-intervention intake of breakfast | 5.54 (1.61) | 5.86 (1.66)
  Two-week Post-intervention Weekly intake of breakfast | 5.77 (1.64) | 5.93 (.92)
  Two-week Post-intervention Weekly intake of family dinner | 4.85 (1.72) | 4.5 (2.03)
Statistical Analysis 1: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child weekly intake of breakfast. It is an independent samples t test. It is testing the null hypothesis that the mean change in child breakfast meals per week from baseline to two-week follow up does not differ between conditions; Test type: Superiority; p = .777, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = -.159, 95% CI 2-sided [-1.33 to 1.01], Standard Error of Mean .55
Statistical Analysis 2: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child intake of family dinners. It is an independent samples t test. It is testing the null hypothesis that the mean change in child family dinners per week from baseline to two-week follow up does not differ between conditions; Test type: Superiority; p = .329, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = -.736, 95% CI 2-sided [-2.26 to .79], Standard Error of Mean .74

10. Secondary Outcome: Change in Screen Time and Activity Behavior
Description: Parents reported on their child's activity behavior of the previous week with two different items asking parents to report the average number of hours per day the child engaged in screen time and physical activity, on a scale from 1 to 5, with 1 = none; 2 = less than 1 hour per day; 3 = 1 to 2 hours per day; 4 = 3 to 4 hours per day; 5 = more than 4 hours per day.
Time Frame: Immediately pre intervention/control and at 2 week follow-up
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video | Virtual Reality
Number analyzed (Participants) | 13 | 14
units on a scale
  Pre-intervention screen time | 4.31 (.88) | 4.11 (1.02)
  Pre-intervention active hours | 2.35 (.72) | 2.89 (.66)
  Two-week Post-intervention screen time | 3.35 (1.05) | 3.61 (1.20)
  Two-week Post-intervention active hours | 2.54 (.80) | 2.96 (.46)
Statistical Analysis 1: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child screentime. It is an independent samples t test. It is testing the null hypothesis that the mean change in child screentime per week from baseline to two-week follow up does not differ between conditions; Test type: Superiority; p = .086, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = .46, 95% CI 2-sided [-0.07 to .99], Standard Error of Mean .26
Statistical Analysis 2: Comparison: Video vs Virtual Reality; This analysis is for the outcome: Change in child active hours. It is an independent samples t test. It is testing the null hypothesis that the mean change in child active hours per week from baseline to two-week follow up does not differ between conditions; Test type: Superiority; p = .64, t-test, 2 sided — A priori threshold for statistical significance set at p<.05; Degrees of freedom = 25; Mean Difference (Net) = -.12, 95% CI 2-sided [-.64 to .40], Standard Error of Mean .25

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and other (non-serious adverse) events were not assessed for the study.
Arm/Group | Video | Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT04845568/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT04845568/ICF_001.pdf